CLINICAL TRIAL: NCT03434132
Title: Open Versus Robot Assisted Radical Cystectomy With Totally Intracorporeal Urinary Diversion. Single Centre Prospective Randomized Trial.
Brief Title: Open Versus Robot Assisted Radical Cystectomy With Totally Intracorporeal Urinary Diversion.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Ministero della Salute, Italy (Other)
Responsible Party: Principal Investigator, Giuseppe SImone, MD, PhD, COnsultant Urologist, Regina Elena Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GR2016-02364306
Record Dates: First submitted 2018-01-26; First posted 2018-02-15 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Bladder Cancer
Keywords: Open Radical Cystectomy; Robotic Radical cystectomy; Intracorporeal urinary diversion; Prospective randdomized trial
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Radical Cystectomy (Active Comparator): Open Radical Cystectomy, pelvic lymph node dissection, urinary diversion (neobladder or ileal conduit)
  Interventions: Procedure: Open or robotic radical cystectomy
- Robot assisted radical cystectomy (Experimental): Robot assisted radical cystectomy, pelvic lymph node dissection, intracorporeal urinary diversion (neobladder or ileal conduit)
  Interventions: Procedure: Open or robotic radical cystectomy

INTERVENTIONS:
Procedure: Open or robotic radical cystectomy — ORC and orthotopic ileal neobladder is performed as previously described. A separate package PLND is performed as in open as in robotic surgery. RARC is performed replicating open surgical procedure.
  The orthotopic ileal neobladder model used is the 'vescica ileale padovana' as previously described. An ileal segment, approximately 42 cm long, is chosen at a minimum distance of 20cm far from ileo-cecal valve. A latero-lateral ileal anastomosis is performed with staplers to restore bowel continuity.
  For ileal conduit, a 20cm ileal segment (approximately 20 cm long) at a minimum distance of 20 cm from ileo-cecal valve is isolated and transected with staplers. Bowel continuity is restored as previously described. The ileal loop on its distal edge is extracted through abdomen wall at the previously identified stoma point and fixed to abdomen fascia. The ureters are spatulated and a latero-lateral anastomosis according to Wallace 1 technique is performed.

SUMMARY:
This prospective randomized study is designed to provide high level of evidence supporting superiority of robot assisted (RA) versus open (O) radical cystectomy (RC). The primary endpoint is a 50% reduction of transfusion rate, several perioperative outcomes potentially linked to a reduced invasiveness are considered as secondary endpoints. Investigators hypothesis is that the reduced invasiveness of RARC might turn into a higher adherence to enhanced recovery after surgery (ERAS) protocols (early bowel recovery, reduced need for painkillers and insertion of nasogastric tube) and consequently to shorter hospital stay and to faster return to daily activities. These data will be taken into account in a matched cost analysis between arms. Secondary aims include a between arm matched comparison of perioperative complications, oncologic outcomes (2-yr disease free survival is an accepted surrogate of long term oncologic effectiveness of RC) and functional outcomes (daytime and nighttime continence).

DETAILED DESCRIPTION:
Despite encouraging data deriving from colorectal surgery, evidences in favor to ERAS protocols following RARC are poor. Moreover, according to a recent survey of surgeons with a specialist interest in RC, the adherence to ERAS protocols is <20% [1].

Retrospective and preliminary data from the robotic consortium have supported oncologic effectiveness of RARC; however in the only prospective randomized trial comparing RARC and ORC urinary diversions were performed extracorporeally, potentially impairing the benefits of minimally invasive surgery [2].

Robot assisted radical cystectomy (RARC) has the aim of providing adequate cancer control while minimizing invasiveness of open radical cystectomy (ORC). The primary end-point of this trial is to demonstrate a reduction of perioperative transfusion rate in RARC arm by 50% compared to ORC arm.

ERAS protocols may significantly contribute to shortening length of hospital stay, a key outcome in this clinical setting of patients receiving RC, being the mean length of hospital stay around 14 days in Italy. Investigators' hypothesis is that the reduced invasiveness of RARC might contribute to an increased adoption of ERAS protocols (reduced need for reinsertion of nasogastric tube, shorter time to first flatus, to mobilization, to regular diet and finally shorter duration of hospital stay).

Assessment of oncologic outcomes of RARC, although not the primary endpoint of the present study, is certainly an outcome of interest. The expected duration of enrollment (18 mo) should provide 2-yr oncologic outcomes for about 66% of patients. Two-year recurrence free survival has been reported as a valid surrogate marker of long term oncologic survival after RC.

Specific Aim 1:To demonstrate superiority of RARC versus ORC in terms of 50% reduction of perioperative transfusion rates.

Specific Aim 2:

To evaluate invasiveness of both surgical approaches by assessing the adherence to ERAS protocols in both and the incidence of perioperative and 30-d, 90d, 180d complications, readmission rates (30d, 90d). Cost analysis will assess the potential impact of shorter hospital stay on overall costs of robotic procedures.

Specific Aim 3:

To assess quality of life at 6-mo, 12-mo and 24-mo follow-up evaluation and to perform a matched comparison of oncologic and functional outcomes between two arms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with muscle invasive high grade urothelial carcinoma (and variant histologies) of the bladder or high grade non muscle invasive BCG recurrent/refractory disease.

Exclusion Criteria:

* Cystectomy without curative intent (palliative, salvage).
* Patients unfit for robotic cystectomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants requiring perioperative transfusions. | 30 days
  50% reduction of perioperative transfusion rates in robotic arm.

SECONDARY OUTCOMES:
Number of participants requiring insertion of nasogastric tube | 30 days
  Comparison between open and robotic arms.
Incidence of Clavien grade 1-2 perioperative complications at 30-d evaluation. | 30 days
  Comparison between open and robotic arms.
Incidence of Clavien grade 1-2 perioperative complications at 90-d evaluation. | 90 days
  Comparison between open and robotic arms.
Incidence of Clavien grade 1-2 perioperative complications at 180-d evaluation. | 180 days
  Comparison between open and robotic arms.
Incidence of patients requiring readmission. | 90 days
  Comparison between open and robotic arms.
Cost analysis. | 30 days
  Comparison between open and robotic arms.

OTHER OUTCOMES:
Assessment of quality of life at 6-mo follow-up with self-administered EORTC QLQ-BLM30 questionnaire | 6 months
  Comparison between open and robotic arms.
Assessment of quality of life at 6-mo follow-up with self-administered EORTC QLQ-C30 questionnaire | 6 months
  Comparison between open and robotic arms.
Assessment of quality of life at 12-mo follow-up with self-administered EORTC QLQ-BLM30 questionnaire | 12 months
  Comparison between open and robotic arms.
Assessment of quality of life at 12-mo follow-up with self-administered EORTC QLQ-C30 questionnaire | 12 months
  Comparison between open and robotic arms.
Assessment of quality of life at 24-mo follow-up with self-administered EORTC QLQ-BLM30 questionnaire | 24 months
  Comparison between open and robotic arms.
Assessment of quality of life at 24-mo follow-up with self-administered EORTC QLQ-C30 questionnaire | 24 months
  Comparison between open and robotic arms.
Disease free survival | 24 months
  Comparison between open and robitic arms
Cancer specific survival | 24 months
  Comparison between open and robitic arms
Overall survival | 24 months
  Comparison between open and robitic arms
Assessment of urinary continence with pad test. | 12 months
  Comparison between open and robotic arms
Assessment of urinary continence with pad test. | 24 months
  Comparison between open and robotic arms

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Simone, PhD, Principal Investigator — "Regina Elena" National Cancer Institute, Dept of Urology
Locations (1):
- Regina Elena NCI, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mastroianni R, Tuderti G, Anceschi U, Bove AM, Brassetti A, Ferriero M, Zampa A, Giannarelli D, Guaglianone S, Gallucci M, Simone G. Comparison of Patient-reported Health-related Quality of Life Between Open Radical Cystectomy and Robot-assisted Radical Cystectomy with Intracorporeal Urinary Diversion: Interim Analysis of a Randomised Controlled Trial. Eur Urol Focus. 2022 Mar;8(2):465-471. doi: 10.1016/j.euf.2021.03.002. Epub 2021 Mar 10. PMID 33712389